CLINICAL TRIAL: NCT02674282
Title: Maximum Oxygen Uptake in ACL-injured Professional Soccer Players
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Adriano Marques de Almeida, Medical Doctor, University of Sao Paulo
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IOT983
Record Dates: First submitted 2016-02-01; First posted 2016-02-04 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Anterior Cruciate Ligament Injury
Keywords: anterior cruciate ligament reconstruction; anterior cruciate ligament; sports medicine; soccer; maximum oxygen uptake; return to play
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ACL-injured (Experimental): ACL injured professional soccer players submitted to ACL reconstruction.
  Interventions: Procedure: ACL reconstruction
- Control (No Intervention): Healthy professional soccer players

INTERVENTIONS:
Procedure: ACL reconstruction — ACL reconstruction with hamstrings autograft.
  Arms: ACL-injured

SUMMARY:
Our purpose is to evaluate maximum oxygen uptake (VO2max) in ACL-injured professional soccer players and after a six-month period of post-operative rehabilitation, compared to a control group of healthy professional soccer players.

DETAILED DESCRIPTION:
The anterior cruciate ligament (ACL) rupture is considered a major injury and may affect the career of professional soccer players. Surgical ACL reconstruction is often required to treat the resulting knee instability. Although ACL reconstruction is considered a successful procedure in restoring knee stability, literature shows that only 55% of the participants return to competitive sports participation after surgery. Soccer players need technical, tactical and physical skills to succeed, such as good knee function and aerobic capacity. Our purpose is to evaluate maximum oxygen uptake (VO2max) in ACL-injured professional soccer players and after a six-month period of post-operative rehabilitation, compared to a control group of healthy professional soccer players.

ELIGIBILITY:
Inclusion Criteria:

* ACL injury
* professional soccer player
* adult
* male

Exclusion Criteria:

* Multiple ligament injury
* knee effusion
* unable to perform the examination on the treadmill
* ACL reconstruction failure
* reoperation due to any cause during the follow-up period
* goalkeeper

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-01; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Maximum oxygen uptake | 6 months
  Ergospirometric evaluation of maximum oxygen uptake running on a treadmill

SECONDARY OUTCOMES:
Running economy | 6 months
  Running economy evaluated on a treadmill
Body composition | 6 months
  Evaluation of body composition with bioimpedance
Isokinetic strength | 6 months
  Quadriceps and hamstrings isokinetic strength evaluation
Knee function | 6 months
  Knee function Lysholm and International Knee Documentation Committee questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Arnaldo J Hernandez, MD, PhD, Study Director — Department of Orthopedics and Traumatology
Locations (1):
- Instituto de Ortopedia e Traumatologia - HCFMUSP, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ardern CL, Taylor NF, Feller JA, Webster KE. Fifty-five per cent return to competitive sport following anterior cruciate ligament reconstruction surgery: an updated systematic review and meta-analysis including aspects of physical functioning and contextual factors. Br J Sports Med. 2014 Nov;48(21):1543-52. doi: 10.1136/bjsports-2013-093398. Epub 2014 Aug 25. PMID 25157180
- [Background] Helgerud J, Engen LC, Wisloff U, Hoff J. Aerobic endurance training improves soccer performance. Med Sci Sports Exerc. 2001 Nov;33(11):1925-31. doi: 10.1097/00005768-200111000-00019. PMID 11689745
- [Background] Stolen T, Chamari K, Castagna C, Wisloff U. Physiology of soccer: an update. Sports Med. 2005;35(6):501-36. doi: 10.2165/00007256-200535060-00004. PMID 15974635